CLINICAL TRIAL: NCT00684320
Title: Attention Disengagement Training for Social Phobia
Acronym: SPAttn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nader Amir, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34MH073004-03 (NIH); R34MH073004-03 (NIH)
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Information Processing; Attention Bias
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 Placebo Condition (PC) (Active Comparator): The placebo, group will complete the PC procedure, which is identical to the ADT procedure except that during the presentation of the trials where a disgust or angry face is present, the probe will appear with equal frequency in the position of disgust or angry and neutral face. Thus, disgust, angry nor neutral face will have signal value regarding the position of the probe.
  Interventions: Behavioral: Placebo Condition
- 1 Attention Disengagement Training (ADT) (Experimental): Those assigned to ADT condition will receive a computer delivered attention retraining protocol designed to enhance attention disengagement from socially threatening stimuli. The ADT protocol includes eight 30-min sessions delivered over a 6-week period (i.e., bi-weekly sessions). During each session, participants will see 320 trials that consist of the various combinations of probe type (E or F) probe position (top or bottom), and emotion type (Neutral, Disgust, Anger). 256 trials will include one neutral face and one disgust face or one angry face: 2 (probe type) X 2 (probe position) X 16 (person) X 4 (repetitions). On trials where participants see one neutral face and one disgust or angry face (i.e., 80% of the trials), the probe will always follow the neutral face.
  Interventions: Behavioral: Attention Disengagement Training (ADT)

INTERVENTIONS:
Behavioral: Attention Disengagement Training (ADT) — Those assigned to ADT condition will receive a computer delivered attention retraining protocol designed to enhance attention disengagement from socially threatening stimuli. The ADT protocol includes eight 30-min sessions delivered over a 6-week period (i.e., bi-weekly sessions). During each session, participants will see 320 trials that consist of the various combinations of probe type (E or F) probe position (top or bottom), and emotion type (Neutral, Disgust, Anger). 256 trials will include one neutral face and one disgust face or one angry face: 2 (probe type) X 2 (probe position) X 16 (person) X 4 (repetitions). On trials where participants see one neutral face and one disgust or angry face (i.e., 80% of the trials), the probe will always follow the neutral face.
  Arms: 1 Attention Disengagement Training (ADT)
Behavioral: Placebo Condition — The placebo condition (PC) will be identical to the AMP condition except that during the presentation of the trials where a threat picture is present, the probe will appear with equal frequency in the position of threat and neutral pictures. Thus, neither threat nor neutral pictures have signal value with regard to the position of the probe.
  Arms: 2 Placebo Condition (PC)

SUMMARY:
Generalized Social Phobia is characterized by severe social anxiety that leads to functional impairment (Schneider et al., 1992). Despite its high prevalence, many individuals do not receive treatment or are unresponsive to current therapies. Thus there is a clear need to continue to develop highly effective and efficient treatments for social phobia. This three year project aims to test a computerized treatment for social phobia in a double-blind, placebo-controlled study designed to modify attention biases that may maintain anxiety.

DETAILED DESCRIPTION:
Generalized Social Phobia (GSP) is characterized by severe social anxiety that leads to functional impairment (Schneider, et al., 1992). The prevalence of GSP is 13.3% (lifetime, Kessler, et al., 1994), ranking third among all psychiatric disorders. Despite its high prevalence, over 30% of individuals with social anxiety who need treatment do not receive treatment for a variety of reasons (e.g., afraid of what others might think, Olfson, et al., 2000). Additionally, 40% of individuals who present for treatment do not respond (39% Heimberg, et al., 1998; 42%, Liebowitz et al., 2005). Thus, there is a clear need to develop highly effective and efficient treatment procedures for social phobia. This three-year proposal aims to test a computerized treatment for social anxiety in a double-blind, placebo-controlled study. Specifically, research suggests that individuals with social phobia direct their attention toward socially-relevant negative information. Therefore, the treatment will focus on changing this attention bias and thereby alleviate symptoms of social anxiety. We present the results of a pilot study (n=26) in treatment seeking socially phobic individuals demonstrating the effectiveness of the treatment. A larger study would allow us to test the treatment and perhaps modify its component to increase its efficacy. The preliminary results of the pilot are encouraging. In brief, our intervention was effective in: a) changing biased attention in socially anxious individuals, b) generalizing this change in disengagement of attention from threat to other measures of attention disengagement, c) reduce symptoms of social anxiety as assessed by an independent rater, d) maintain a high rate of compliance (0% drop out in the pilot study), and e) maintain its effects in follow-up assessment up to one year. This efficient and efficacious techniques for changing attention bias in social phobia can provide a cost-effective and easy to administer treatment that is grounded in basic cognitive science and may help reduce suffering in individuals with GSP. We will test two hypotheses in this proposal. 1) Individuals with GSP completing the Attention Disengagement Training (ADT) will show a larger reduction in their symptoms compared to the placebo group on an interviewer measure of social anxiety (Liebowitz Social Anxiety Scale, LSAS). 2) Individuals with GSP completing ADT will show a larger reduction in their self-report of social anxiety symptoms compared to the placebo group

ELIGIBILITY:
Inclusion Criteria:

* Principle DSM-IV-TR (APA, 2000) Diagnosis of social phobia - Generalized Type (GSP)

Exclusion Criteria:

* No change in medication type or dosage twelve weeks prior to initiating treatment
* No current psychotherapy
* No evidence of suicidal intent
* No evidence of substance abuse in the last 6 months
* No evidence of current or past schizophrenia, bipolar disorder, or organic mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Amir, Ph.D., Principal Investigator — SDSU/UCSD
Locations (1):
- San Diego State University, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2 Placebo Condition (PC) | 1 Attention Disengagement Training (ADT)
Started | 26 | 22
Completed | 22 | 22
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Placebo Condition (PC) | 1 Attention Disengagement Training (ADT) | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 48
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  male | 11 | 8 | 19
  female | 13 | 14 | 27
  unreported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Liebowitz Social Anxiety Scale (LSAS)
Description: Our primary outcome measure was the clinician-administered LSAS (Liebowitz, 1987), a 24-item scale that provides separate scores for fear and avoidance of social interaction and performance situations. LSAS scores range from 0 to 144. The LSAS has strong psychometric properties (Heimberg et al., 1999) and is arguably the gold-standard outcome measure in treatment research in SAD (e.g., Clark et al., 2006; Heimberg et al., 1998). Higher scores indicate more severe symptoms
Time Frame: Pre-Treatment, Post-Treatment (6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2 Placebo Condition (PC) | 1 Attention Disengagement Training (ADT)
Number analyzed (Participants) | 22 | 22
units on a scale
  Pre-Treatment | 68.1 (16.7) | 74.5 (16.6)
  Post-Treatment | 60.0 (18.2) | 46.1 (16.6)

2. Secondary Outcome: Social Phobia and Anxiety Inventory
Description: Our primary self-report outcome measure was the Social Phobia and Anxiety Inventory (SPAI; Turner, Beidel, Dancu, & Stanley, 1989), which consists of 45 items assessing the cognitive, behavioral, and somatic dimensions of SP. SPAI scores range from 45 to 315, with higher scores indicating more severe symptoms. This measure has strong psychometric properties (Turner et al., 1989) and has been widely used in previous treatment outcome research in SP (e.g., Clark et al., 2006).
Time Frame: Pre-Treatment, Post-Treatment (after 4 weeks of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2 Placebo Condition (PC) | 1 Attention Disengagement Training (ADT)
Number analyzed (Participants) | 22 | 22
units on a scale
  Pre-Treatment | 126.7 (20.9) | 132.3 (17.3)
  Post-Treatment | 109.0 (30.9) | 99.1 (30.8)

ADVERSE EVENTS:
Arm/Group | 2 Placebo Condition (PC) | 1 Attention Disengagement Training (ADT)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes